CLINICAL TRIAL: NCT05695547
Title: Non-inferiority of Virtual Reality Augmented Education in Patients Undergoing Coronary Angiography
Brief Title: VR Education in Patients Undergoing Coronary Angiography
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Adela Drozdova (Other)
Responsible Party: Sponsor-Investigator, Adela Drozdova, PI, Nemocnice AGEL Trinec-Podlesi a.s.
Organization: Nemocnice AGEL Trinec-Podlesi a.s. (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AGELTrinecPodlesi VR2
Record Dates: First submitted 2023-01-05; First posted 2023-01-25 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Coronary Arteriosclerosis
Keywords: Virtual Reality; Education
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard education (No Intervention): Patients will be educated about the procedure in a standard way by a doctor and a nurse
- VR Education (Experimental): Patients will be educated with the use of virtual reality
  Interventions: Other: VR educational video

INTERVENTIONS:
Other: VR educational video — Patients will be educated with our specifically made VR video in the settings of our hospital to make patients more familliar with the spaces and to explain them the procedure.
  Arms: VR Education

SUMMARY:
The aim of this study is to compare standard education with VR augmented education in patients undergoing selective coronary angiography.

DETAILED DESCRIPTION:
The aim of this study is to compare standard education (doctor and nurse led) with Virtual Reality (VR) augmented education in patients prior toa selective coronary angiography. A 360° education video was prepared in the operating theatre and other areas of the hospital to make patients more comfortable with these unfamilliar places. The procedure was explained in details by a doctor and animations were used to help them to visualise the procedure. Risks and complications of the procedure were highlited along with the precautionary measures the patient need to take after the procedure.

Patients coming into the One-Day Cardilogy Unit of Podlesi Hospital will be randomised into 2 groups: Standard education and VR augmented education. The VR group will be then educated using VR and will be given an opportunity to ask a physician more questions if needed. Patients will then fill in forms to assess their experience, feelings and knowledge about the procedure. Data will be then collected to assess if VR could facilitate patients' education. The investigators believe it could be a useful tool to save time of doctors and nurses which is becoming more and more precious and expensive.

ELIGIBILITY:
Inclusion Criteria:

* Patients with indication for undergoing coronary angiography

Exclusion Criteria:

* Visual impairment

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-01-25 (Estimated); Primary Completion 2024-01-05 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Quality of VR augmented eduacation assessed by a questionaire | 18 months
  A questionaire with questions assessing patients' personal experience and knowledge of the procedure was prepared.
  This will be collected and compared to patients with a standard education.

IPD SHARING:
Plan to Share IPD: Undecided
general demographic data